CLINICAL TRIAL: NCT00004817
Title: Phase III Double Blind Trial of Valproate Sodium for Prophylaxis of Post Traumatic Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Harborview Injury Prevention and Research Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/12249; UW-19643
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Post-Traumatic Seizure Disorder; Head Injuries
Keywords: neurologic and psychiatric disorders; rare disease; seizures
MeSH Terms: conditions — Epilepsy, Post-Traumatic; Craniocerebral Trauma; Neurologic Manifestations; Mental Disorders; Rare Diseases; Seizures | interventions — Phenytoin; Valproic Acid

INTERVENTIONS:
Drug: phenytoin
Drug: valproate sodium

SUMMARY:
OBJECTIVES: I. Determine whether treating head injured patients with valproate sodium will reduce the risk of developing seizures as a result of the head injury.

II. Determine the safety of valproate, the appropriate dose, and the effect valproate may have on the recovery of the brain's ability to compute numbers, solve problems, remember information, and control the movement of limbs after head injury.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind trial involving 3 treatment groups.

On day 1, controls receive phenytoin IV over 1 hour. On days 2 through 7, controls receive 2 doses each of phenytoin and placebo daily, intravenously. From day 8 through 6 months, controls receive placebo IV 4 times daily, then placebo tablets are administered.

On day 1, the experimental group receives a loading dose of valproate sodium intravenously over 1 hour within 24 hours of injury. Then, patients are divided into 2 subgroups.

From day 2 through 1 month, one group of patients receives valproate IV 4 times daily over 1 hour until tablets are tolerated. Patients receive placebo tablets by mouth 4 times daily from month 2 through month 6.

On day 2, the other group of patients receives valproate IV 4 times daily and continues for 6 months until tablets (same dose) are tolerated.

If patients remain seizure free between day 8 and 6 months, the number of valproate or placebo tablets are tapered over 1 week.

Each patient receives a full neuropsychological and psychosocial examination at 1, 6, and 12 months after injury.

Untreated observation of patients continues until 2 years after injury.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Any patient developing the following conditions within 24 hour postinjury:

* Cortical contusion
* Depressed skull fracture
* Subdural hematoma
* Epidural hematoma
* Intracerebral hematoma
* Penetrating head wound
* Seizures occurring subsequent to head injury

--Prior/Concurrent Therapy--

* No antiseizure medication prior to injury or between the injury and study drug loading
* Surgery: No prior neurosurgical operation for which the skull and dura mater were opened

--Patient Characteristics--

* Age: 14 and over
* Hematopoietic: No abnormal coagulation profile
* Hepatic: No history of chronic or alcoholic liver disease Adequate liver function as indicated by ALT less than 1.5 times the upper limit of normal
* Other: Not pregnant No injuries greater than 24 hours old No history of seizures prior to injury No prior history of significant head injury or neurological condition requiring medical attention

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 385
Dates: Start 1991-02

CONTACTS AND LOCATIONS:
Overall Officials: H. Richard Winn, Study Chair — Harborview Injury Prevention and Research Center